CLINICAL TRIAL: NCT02152371
Title: A Randomized, Double-Blind Trial Comparing the Effect of Dulaglutide 1.5 mg With Placebo on Glycemic Control in Patients With Type 2 Diabetes on Basal Insulin Glargine
Brief Title: A Study of Dulaglutide (LY2189265) in Participants With Type II Diabetes
Acronym: AWARD-9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13195; H9X-MC-GBDI (Other: Eli Lilly and Company); 2012-004229-25 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin Glargine; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dulaglutide + Insulin Glargine (Experimental): 1.5 milligrams (mg) dulaglutide administered subcutaneously (SQ) once weekly for 28 weeks. Titrated insulin glargine administered SQ once daily for 28 weeks. Participants who are taking metformin should remain on stable doses.
  Interventions: Drug: Dulaglutide; Drug: Insulin Glargine; Drug: Metformin
- Placebo + Insulin Glargine (Placebo Comparator): Placebo administered SQ once weekly for 28 weeks. Titrated insulin glargine administered SQ once daily for 28 weeks. Participants who are taking metformin should remain on stable doses.
  Interventions: Drug: Placebo; Drug: Insulin Glargine; Drug: Metformin

INTERVENTIONS:
Drug: Dulaglutide — Administered SQ
  Other Names: LY2189265
  Arms: Dulaglutide + Insulin Glargine
Drug: Placebo — Administered SQ
  Arms: Placebo + Insulin Glargine
Drug: Insulin Glargine — Administered SQ
Drug: Metformin — Administered orally

SUMMARY:
The main purpose of this study is to evaluate the use of the study drug known as dulaglutide in participants with type II diabetes who are taking once-daily insulin glargine. The study will last about 31 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (based on the World Health Organization's [WHO] diagnostic criteria)
* Have been treated with basal insulin glargine once daily with or without metformin for at least 3 months prior to screening
* Doses of once daily insulin glargine and metformin (if taken) must be stable during the 3-month period prior to screening. Doses of metformin are considered stable if all prescribed doses during this period are in the range between the minimum required dose (≥1500 mg/day) and the maximum approved dose per the locally-approved label
* Have an HbA1c value ≥7.0% and ≤10.5% as assessed by the central laboratory at screening
* Require further insulin glargine dose increase at week 3 per the treat-to-target (TTT) algorithm based on the SMPG data collected during the prior week
* Have stable weight (±5%) ≥3 months prior to screening
* Have body mass index (BMI) ≤45 kilograms per square meter (kg/m^2) at screening
* Are able and willing to administer once weekly randomized therapy
* Are females of childbearing potential who must:

  * Test negative for pregnancy at screening, based on a serum pregnancy test
  * Agree to use a reliable method of birth control
  * Not be breastfeeding

Exclusion Criteria:

* Have been treated with ANY other antihyperglycemia regimen, other than basal insulin glargine once daily with or without metformin, within the 3 months prior to screening or between screening and week 3
* Have a history of ≥1 episode of ketoacidosis or hyperosmolar state/coma
* Have a history of hypoglycemia unawareness within the 6 months prior to screening
* Have been treated with drugs that promote weight loss within the 3 months prior to screening or between screening and week 3
* Are receiving chronic (>14 days) systemic glucocorticoid therapy or have received such therapy within the 4 weeks prior to screening or between screening and week 3
* Have had any of the following cardiovascular conditions within the 2 months prior to screening: acute myocardial infarction (MI), New York Heart Association (NYHA) Class III or Class IV heart failure, or cerebrovascular accident (stroke)
* Have a known clinically significant gastric emptying abnormality or have undergone gastric bypass surgery or restrictive bariatric surgery
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or alanine aminotransferase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory
* Have a history of chronic pancreatitis or acute idiopathic pancreatitis, or were diagnosed with any type of acute pancreatitis within the 3 months prior to screening
* Have an estimated glomerular filtration rate (eGFR) <30 milliliters/minute/1.73 square meter (mL/min/m^2), calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation, as determined by the central laboratory; for participants on metformin, have renal disease or renal dysfunction (for example, a serum creatinine ≥1.5 mg/deciliter [dL] [male] or ≥1.4 mg/dL [female] or eGFR [CKD-EPI] <60 mL/min/1.73 m^2)
* Have evidence of a significant, uncontrolled endocrine abnormality
* Have any self or family history of type 2A or type 2B multiple endocrine neoplasia (MEN 2A or 2B) in the absence of known C-cell hyperplasia
* Have any self or family history of medullary C-cell hyperplasia, focal hyperplasia, or carcinoma (including sporadic, familial, or part of MEN 2A or 2B syndrome)
* Have serum calcitonin ≥20 picograms/mL, as determined by the central laboratory
* Have evidence of a significant, active autoimmune abnormality
* Have any other condition not listed in this section that is a contraindication for use of insulin glargine, or, for participants using metformin, have a condition that is a contraindication for the use of metformin and would require metformin discontinuation per label
* Have a history of transplanted organ
* Have a history of active or untreated malignancy, or are in remission from a clinically significant malignancy during the 5 years prior to screening
* Have a history of any other condition which, in the opinion of the investigator, may preclude the participants from following and completing the protocol
* Have any hematologic condition that may interfere with HbA1c measurement (eg, hemolytic anemias, sickle-cell disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (13):
  - Valley Endocrine, Fresno, Fresno, California
  - Mills-Peninsula Diabetes Research Insitute, San Mateo, California
  - University Clinical Investigators, Inc., Tustin, California
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Northwest Endo Diabetes Research, LLC, Arlington Heights, Illinois
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - AB Clinical Trials, Las Vegas, Nevada
  - SHS Clinical Research Group, Toms River, New Jersey
  - Bland Clinic, PA, Greensboro, North Carolina
  - PMG Research of Knoxville, Knoxville, Tennessee
  - Rainier Clinical Research Center, Renton, Washington
  - Polyclinic, Seattle, Washington
- Czechia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beroun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandys Nad Labem-Stara Bolesl
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., České Budějovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krnov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Hungary (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagykanizsa
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Puerto Rico (6):
  - Centro de Endocrinologia y Nutricion del Turabo, Caguas
  - Manati Center for Clinical Research Inc, Manatí
  - Ponce School of Medicine CAIMED Center, Ponce
  - Endocrine Lipid Diabetes Research Institute, Ponce
  - GCM Medical Group PSC, San Juan
  - American Telemedicine Center, San Juan
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cadiz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mortimer, Berks
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leicester, Leicestershire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guildford, Surrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Swansea, Wales

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Pantalone KM, Patel H, Yu M, Fernandez Lando L. Dulaglutide 1.5 mg as an add-on option for patients uncontrolled on insulin: Subgroup analysis by age, duration of diabetes and baseline glycated haemoglobin concentration. Diabetes Obes Metab. 2018 Jun;20(6):1461-1469. doi: 10.1111/dom.13252. Epub 2018 Mar 23. PMID 29430801
- [Derived] Yu M, Brunt KV, Milicevic Z, Varnado O, Boye KS. Patient-reported Outcomes in Patients with Type 2 Diabetes Treated with Dulaglutide Added to Titrated Insulin Glargine (AWARD-9). Clin Ther. 2017 Nov;39(11):2284-2295. doi: 10.1016/j.clinthera.2017.10.002. Epub 2017 Oct 27. PMID 29110972

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible participants entered a 2-week lead-in period. Only those participants who required further up-titration of the insulin glargine dose per treat-to-target (TTT) algorithm were randomized to one of two treatment groups.
Period: Overall Study
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Started | 150 | 150
Received at Least 1 Dose of Study Drug. | 150 | 150
Completed | 138 | 134
Not Completed | 12 | 16
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Reason Not Given | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.47) | 60.6 (10.07) | 60.4 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 62 | 127
  Male | 85 | 88 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 25 | 51
  Not Hispanic or Latino | 104 | 104 | 208
  Unknown or Not Reported | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 5 | 6 | 11
  White | 143 | 138 | 281
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czech Republic | 25 | 27 | 52
  Puerto Rico | 12 | 16 | 28
  Hungary | 37 | 35 | 72
  United States | 32 | 29 | 61
  Italy | 13 | 15 | 28
  United Kingdom | 2 | 2 | 4
  Spain | 29 | 26 | 55
Mean Insulin Glargine Dose [Mean (Standard Deviation); unit: Units (U)] | 40.71 (23.12) | 36.59 (21.46) | 38.65 (22.37)
Metformin Use at Baseline [Number; unit: participants]
  Treated with Metformin | 134 | 131 | 265
  Not Treated with Metformin | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 28 Weeks in Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least-squares (LS) mean and standard error (SE) changes from baseline in HbA1c at 28 weeks were measured using mixed model regression and restricted maximum likelihood (REML) with treatment, pooled country, visit, and treatment-by -visit interaction as fixed effects, baseline as covariate, and participant as a random effect.
Time Frame: Baseline, 28 Weeks
Population: All participants who received at least one dose of study drug and had evaluable baseline and post- baseline HbA1c.
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of change | -1.44 (0.09) | -0.67 (0.09)
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Mixed Model for Repeated Measures (MMRM); LS Means Diff = -0.77, 95% CI 2-sided [-0.97 to -0.56], Standard Error of Mean 0.10

2. Secondary Outcome: Change From Baseline to 28 Weeks in Fasting Serum Glucose (FSG)
Description: FSG is a test to determine glucose levels after an overnight fast. LS means FSG change from baseline to primary endpoint at week 28 was calculated using a mixed effects model for repeated measures (MMRM) analysis adjusted by treatment, country, metformin use, week, treatment-by-week interaction, and baseline FSG as covariate.
Time Frame: Baseline, 28 Weeks
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline FSG data.
Measure: Least Squares Mean (Standard Error); unit: milligram per deciliter (mg/dL)
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
milligram per deciliter (mg/dL) | -44.63 (4.16) | -27.90 (4.08)
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -16.73, 95% CI 2-sided [-26.02 to -7.44], Standard Error of Mean 4.72

3. Secondary Outcome: Change From Baseline to 28 Weeks in 7-Point Self Monitored Plasma Glucose (SMPG)
Description: The LS means of the 7-point SMPG change from baseline to primary endpoint at week 28 was measured using a MMRM analysis adjusted by treatment, country, metformin use, week, treatment-by-week interaction, and baseline SMPG as covariate.
Time Frame: Baseline, 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had evaluable baseline and post-baseline SMPG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
mg/dL
  Pre-Morning Meal (n=133,129) | -44.03 (2.71) | -35.97 (2.64)
  Morning Meal 2-Hour Postprandial (n=123,119) | -64.16 (4.31) | -46.97 (4.27)
  Pre-Midday Meal (n=133,127) | -40.89 (3.72) | -25.34 (3.62)
  Midday Meal 2-Hour Post Prandial (n=123,117) | -51.13 (4.40) | -32.98 (4.33)
  Pre-Evening Meal (n=133,129) | -43.68 (4.21) | -28.71 (4.07)
  Evening Meal 2-Hour Postprandial (n=126,122) | -48.63 (5.22) | -27.35 (5.16)
  3:00 AM (Morning) (n=124,117) | -39.77 (4.27) | -20.30 (4.23)
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Pre-Morning Meal; Test type: Superiority or Other; p = .007, Mixed Models Analysis; LS Mean Diff = -8.06, 95% CI 2-sided [-13.87 to -2.25], Standard Error of Mean 2.95
Statistical Analysis 2: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Morning Meal 2-Hour Postprandial; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -17.18, 95% CI 2-sided [-25.96 to -8.40], Standard Error of Mean 4.45
Statistical Analysis 3: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Pre-Midday Meal; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -15.55, 95% CI 2-sided [-23.58 to -7.52], Standard Error of Mean 4.08
Statistical Analysis 4: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Midday Meal 2-Hour Postprandial; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -18.15, 95% CI 2-sided [-27.18 to -9.12], Standard Error of Mean 4.58
Statistical Analysis 5: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Pre-Evening Meal; Test type: Superiority or Other; p = .001, Mixed Models Analysis; LS Mean Diff = -14.96, 95% CI 2-sided [-23.93 to -5.99], Standard Error of Mean 4.55
Statistical Analysis 6: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Evening Meal 2-Hour Postprandial; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -21.28, 95% CI 2-sided [-32.46 to -10.10], Standard Error of Mean 5.68
Statistical Analysis 7: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; 3:00AM (Morning); Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Mean Diff = -19.48, 95% CI 2-sided [-28.77 to -10.18], Standard Error of Mean 4.72

4. Secondary Outcome: Change From Baseline to 28 Weeks in Body Weight
Description: LS means of the body weight change from baseline to primary endpoint at week 28 was adjusted by treatment, country, metformin use, week, treatment-by-week interaction, and baseline body weight as covariate, via a MMRM analysis.
Time Frame: Baseline, 28 Weeks
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilogram(kg)
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
kilogram(kg) | -1.91 (0.30) | 0.50 (0.30)
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Mixed Models Analysis; LS Means Difference = -2.41, 95% CI 2-sided [-3.19 to -1.64], Standard Error of Mean 0.39

5. Secondary Outcome: Change From Baseline to 28 Weeks in Daily Mean Insulin Glargine Dose
Description: Least Square (LS) Means of the insulin dose change from baseline to primary endpoint at week 28 was adjusted by treatment, country, metformin use, week, treatment-by-week interaction, and baseline insulin dose as covariate, via a MMRM analysis.
Time Frame: Baseline, 28 Weeks
Population: All participants who one dose of study drug and had evaluable baseline and post-baseline insulin glargine data.
Measure: Least Squares Mean (Standard Error); unit: units (u)
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
units (u) | 12.75 (2.27) | 25.94 (2.30)
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, MMRM; LS Means Diff = -13.19, 95% CI 2-sided [-19.55 to -6.84], Standard Error of Mean 3.21

6. Secondary Outcome: Number of Participants With Investigator Reported and Adjudicated Cardiovascular Events
Description: Cardiovascular (CV) adverse events (AEs) were adjudicated by an independent committee of physicians with cardiology expertise external to the sponsor. Deaths occurring during the study treatment period and nonfatal CV AEs were to be adjudicated. Nonfatal CV events that were to be adjudicated were myocardial infarction; hospitalization for unstable angina; hospitalization for heart failure; coronary interventions (such as coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI); and cerebrovascular events, including cerebrovascular accident (CVA/stroke), and transient ischemic attack (TIA).
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study.
Measure: Number; unit: participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
participants | 3 | 1

7. Secondary Outcome: Percentage of Participants With Self-Reported Events of Hypoglycemia
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of =<3.9 mmol/L), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of =<3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The percentage of participants with self-reported hypoglycemic events is presented.
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants
  Symptomatic | 35.3 | 30.0
  Asymptomatic | 42.7 | 39.3
  Severe | 0.7 | 0.0
  Nocturnal | 28.0 | 28.7
  Probable Symptomatic | 2.7 | 2.0

8. Secondary Outcome: Percentage of Participants Discontinuing the Study Due to Severe, Persistent Hyperglycemia
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants | 0 | 0

9. Secondary Outcome: Number of Participants With Adjudicated Acute Pancreatitis Events
Description: The number of cases of acute pancreatitis confirmed by adjudication. A summary of serious and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
participants | 0 | 0

10. Secondary Outcome: Number of Participants With Thyroid Tumors/Neoplasms (Including C-Cell Hyperplasia)
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
participants | 1 | 0

11. Secondary Outcome: Number of Participants With Dulaglutide Anti-Drug Antibodies
Description: Dulaglutide anti-drug antibodies (ADA) were assessed at baseline, Weeks 12 and 28. A participant was considered to have treatment-emergent (TE) dulaglutide ADAs if the participant had at least 1 titer that was TE relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline, Week 12 and Week 28
Population: All randomized participants who received at least 1 dose of study drug and had at least one post-baseline Dulaglutide ADA test result.
Measure: Number; unit: participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 149 | 149
participants | 0 | 2

12. Secondary Outcome: Percentage of Participants Achieving HbA1c Targets of <7.0% or ≤6.5%
Description: Percentage of participants who achieved HbA1c levels of <7% or ≤6.5% were analyzed using a logistic regression model, controlling for treatment, pre-treatment, baseline HbA1c and country.
Time Frame: 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had a baseline and post-baseline HbA1c data. Last observation carried forward (LOCF) methodology was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants
  HbA1c <= 6.5 | 50.7 | 16.7
  HbA1c < 7.0 | 69.3 | 35.3
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio (OR) = 6.66, 95% CI 2-sided [3.70 to 12.00]
Statistical Analysis 2: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio, log = 5.71, 95% CI 2-sided [3.35 to 9.73]

13. Secondary Outcome: Percentage of Participants Achieving HbA1c Target of <7.0% and Without Weight Gain (<0.1 Kilograms [kg]) at 28 Weeks and Without Documented Symptomatic Hypoglycemia During the Maintenance Period (Weeks 12-28)
Description: Percentage of participants who achieved a target HbA1c target of <7%, without weight gain and without documented symptomatic hypoglycemia at 28 weeks were analyzed using regression model, controlling for treatment, pre-treatment, baseline HbA1c and country.
Time Frame: 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline HbA1c data.Last observation carried forward (LOCF) methodology was used to impute missing post-baseline values.
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants | 40.7 | 16.7
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio (OR) = 4.17, 95% CI 2-sided [2.32 to 7.47]

14. Secondary Outcome: Percentage of Participants Achieving HbA1c Target of <7.0% at 28 Weeks and Without Documented Symptomatic Hypoglycemia During the Maintenance Period (Weeks 12-28)
Description: Percentage of participants achieving target HbA1c of <7.0% at 28 weeks without documented symptomatic hypoglycemia are presented. Documented symptomatic hypoglycemia is defined as any time a participant experienced symptoms and or signs associated with hypoglycemia and had a plasma glucose of <=70 mg/dL.
Time Frame: 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post-baseline HbA1c data. Last observation carried forward (LOCF) methodology was used to impute missing post-baseline values
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants | 52.0 | 28.0
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio (OR) = 3.61, 95% CI 2-sided [2.09 to 6.23]

15. Secondary Outcome: Percentage of Participants Achieving HbA1c Target of <7.0% and Without Weight Gain (<0.1 kg)
Time Frame: 28 Weeks
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
percentage of participants | 52.7 | 20.0
Statistical Analysis 1: Comparison: Dulaglutide + Insulin Glargine vs Placebo + Insulin Glargine; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio (OR) = 5.60, 95% CI 2-sided [3.26 to 9.62]

16. Secondary Outcome: Rate of Hypoglycemic Events up to 28 Weeks
Description: The rate of total hypoglycemic events any type per 30 days is presented. The hypoglycemia rate per 30 days during defined period is calculated by the number of hypoglycemia events within the period/number of days participant at risk within the period*30 days.
Time Frame: Baseline through 28 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: rate of hypoglycemic events per 30 days
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Number analyzed (Participants) | 150 | 150
rate of hypoglycemic events per 30 days | 0.63 (1.24) | 0.70 (1.32)

ADVERSE EVENTS:
Arm/Group | Dulaglutide + Insulin Glargine | Placebo + Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 9/150 | 7/150
Other Adverse Events (participants affected / at risk) | 51/150 | 29/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide + Insulin Glargine (N=150) | Placebo + Insulin Glargine (N=150)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Granulomatous liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dulaglutide + Insulin Glargine (N=150) | Placebo + Insulin Glargine (N=150)
Diarrhoea (Gastrointestinal disorders) | 17 (19) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 18 (23) | 2 (3)
Vomiting (Gastrointestinal disorders) | 9 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 14 (19)
Upper respiratory tract infection (Infections and infestations) | 11 (18) | 10 (10)
Decreased appetite (Metabolism and nutrition disorders) | 10 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days